CLINICAL TRIAL: NCT05793814
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Effects of Consumption of a Limosilactobacillus Supplement on Recurrence of Uncomplicated Symptomatic Urinary Tract Infections (UTI) in Healthy Women During a 6-month Period
Brief Title: Assess the Effects of a Limosilactobacillus Supplement on Recurrence of UTI in Healthy Women During a 6-month Period
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Church & Dwight Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AFCRO-138
Record Dates: First submitted 2023-03-02; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Uncomplicated Symptomatic Urinary Tract Infections
MeSH Terms: interventions — Probiotics; Lacteol

STUDY DESIGN:
Intervention Model Description: A Randomized, Double -Blind, Placebo-Controlled Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Limosilactobacillus Supplement (Experimental): Capsules containing Probiotic taken daily for 6 month
  Interventions: Dietary Supplement: Limosilactobacillus reuteri 3613
- Placebo (Placebo Comparator): Capsules containing Microcrystalline cellulose, magnesium stearate taken Daily for 6 month
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Limosilactobacillus reuteri 3613 — Daily for 6 month
  Other Names: Probiotics, Lactobacillus
  Arms: Experimental: Limosilactobacillus Supplement
Dietary Supplement: Placebo — Daily for 6 month
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to assess the efficacy of the probiotic Limosilactobacillus reuteri 3613 for the decrease or prevent UTI occurrence in women ages 18-65 with a confirmed medical history of recurrent uncomplicated UTIs compared to a Placebo (the study medication without the probiotic)

DETAILED DESCRIPTION:
Adult women with a confirmed medical history of recurrent uncomplicated UTIs meeting all the eligibility criteria will be allocated in two study arms: test and placebo. Approximately 65 subjects per group will be enrolled to assure that approximately 50 subjects in each group complete the study. the study will be conducted in Ireland. The study will last approximately six month for each subject and will consist of 5 visits. The L. reuteri 3613 will be taken daily for 6 months and the frequency of UTIs will be assessed to determine the potential for the probiotic to decrease or prevent UTI occurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to give voluntary, written, informed consent to participate in the trial.
2. Be between 18-65, inclusive.
3. Has a BMI between 18.5 to 40 kg/m2, inclusive.
4. Has a history of recurrent UTIs, defined as ≥ 3 episodes in the past year, of which two were approximately in the past 6 months immediately prior to their screening visit (Visit 1), at the discretion of the investigator. At least one episode must be diagnosed medically and treated by a health care professional, the remaining two may be self-reported.
5. Willing to maintain existing dietary and physical activity patterns throughout the trial period.
6. Willing to comply with the trial protocol and consume the investigational product daily for the duration of the trial.

   -

Exclusion Criteria:

1. Individuals who are on unstable medications (defined as prescribed medications which in the opinion of the investigator may impact the outcomes of the study (defined as prescribed medications for which participant only takes periodically or 'as needed').
2. Individuals with a history of UTIs who have experienced >5 UTIs in the 6 months prior to their Baseline Visit (Week 0).
3. Participants with clinically significant abnormal laboratory results at their screening visit (from urine culture, urinalysis, and safety blood assessments) which, in the opinion of the investigator, would impact the efficacy of the trial or the safety of the participant.
4. Individuals who are pregnant, breastfeeding, or wish to become pregnant during the trial.
5. Individuals currently of childbearing potential, but not using an effective method of contraception
6. Individuals who have taken oral antibiotics (or topical antibiotics in their urogenital area) within the previous 30 days prior to their Baseline Visit (Visit 2).
7. Individuals with a current history of drug abuse (self-report) and/or alcohol abuse (>2 standard alcoholic drinks per day) within the 6 months prior to Baseline Visit (Visit2).
8. Uses tobacco or smoking-related products (including, but not limited to cigarettes, cigars, chewing tobacco, e-cigarettes), and nicotine products (e.g., nicotine gum and/or nicotine patches).
9. Individuals currently consuming an extremely restrictive diet, or in the previous 3 months prior to their Baseline Visit or planning to consume a restrictive diet during the trial.
10. Individuals who are not willing to adhere to dietary/supplement restrictions listed in the trial protocol (refrain from consumption of probiotic supplements, prebiotics, cranberry supplements, and D-mannose supplements; limit consumption of yoghurt, fermented foods, and cranberries to no more than once per week).
11. Individuals with allergies or sensitivities to ingredients that would preclude intake of the investigational products.
12. Participants may not be receiving treatment involving experimental drugs. If the participant has been in a recent experimental trial, these must have been completed not less than 30 days prior to their Screening Visit (Visit 1) for this trial.
13. Individuals that have a significant acute or chronic coexisting illness such as renal diseases (renal failure, nephrolithiasis), anatomical urinary tract abnormalities, intestinal disease, severe uncontrolled metabolic or cardiovascular disease (such as diabetes or hypertension), anticoagulant therapy, cancer, or HIV, or any condition which contraindicates, in the investigator's judgement, entry to the trial.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 130 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of symptomatic UTI | 6 months
  To evaluate in healthy women who experience recurrent UTIs, the effect of 6 months of daily supplementation of the investigational product on incidence rate of symptomatic UTIs.
Proportion of subjects experiencing ≥1 symptomatic UTI | 6 months
  Proportion of participants per product group experiencing ≥1 symptomatic UTI (as determined by urine culture) during the 6-month intervention period (from Baseline Visit [V2] to Final Visit [V5]).

SECONDARY OUTCOMES:
UTI symptom severity | 6 months
  Change in UTI symptom severity of participants with symptomatic UTI between product groups comparing Baseline (Week 0) with scores to scores at V 5 for
Proportion of subjects experiencing different numbers of UTI | 6 months
  Proportion of participants per product group experiencing 0, 1, 2, 3, or more symptomatic UTI during the 6-month intervention period from V2 to Final V5
Total UTI count | 6 months
  Difference in total number of UTIs per group (probiotic treatment compared to placebo group) during the 6-month intervention period from V2 to Final V5
Time for the first UTI | 6 months
  Difference in time from Day 0 to the first UTI occurrence between product groups, during the 6-month intervention period from Day 0 to V5
Vaginal pH change | 6 months
  Change in vaginal pH over time from Visit 2 to Visit 5, between product groups
Quality of Life change | 6 months
  Change in Quality of Life questionnaire using Likert scale over time from Visit 2 to Visit 5, between product groups

OTHER OUTCOMES:
Time for vaginal presence of the probiotic | 6 months
  To evaluate in healthy women who experience recurrent UTIs, the effect of 6 months of daily supplementation of the investigational product on the time it takes for the probiotic to reach the urogenital tract. The probiotic in vaginal samples will be measured visits 2-5.
Vaginal microbiome | 6 months
  Modulation of the vaginal microbiome analyzed using Shotgun metagenomic sequencing from Baseline (Week 0) to Visit 5 (Week 24) compared between groups.
Vaginal presence of the probiotic | 6 months
  To evaluate the proportion of participants with vaginal swabs positive for the probiotic at Baseline (Visit 2) compared to Visit 5 (Week 24, end of intervention) between product groups.
Safety assessment | 6 months
  Occurrence of any Adverse Events (AEs/SAEs).
Tolerability | 6 months
  Vital signs (Blood Pressure, Heart Rate, and Temperature).

CONTACTS AND LOCATIONS:
Locations (1):
- Church &Dwight., Inc, Princeton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided